# Statistical Analysis Plan

# An Open-label, Randomized, Crossover Study in Healthy Volunteers to Compare the Pharmacokinetics of Sotorasib Administered as a 240 mg Tablet or 120 mg Tablets

SAP Status: Final SAP Version: 1.0 SAP Date: 02June2022

Investigational Medicinal Product: Sotorasib (AMG 510)

Protocol Reference: 20210088 Labcorp Drug Development Study: 8471134

Sponsor:

Amgen, Inc.

One Amgen Center Drive

Thousand Oaks, California 91320

**USA** 

Study Sites:

Labcorp Drug Development Clinical

Research Unit

1900 Mason Avenue, Suite 140 Daytona Beach, Florida 32117

**USA** 

Principal Investigators:



Labcorp Drug Development Dallas Clinical

Research Unit

1341 W. Mockingbird Lane, Suite 400E,

Dallas, TX 75247

USA

Labcorp Drug Development Clinical

Research Unit 3402 Kinsman Blvd, Madison, WI, 53704

Information described herein is confidential and may be disclosed only with the express written permission of the sponsor.

NCT Number: NCT05327491
This NCT number has been applied to the document for purposes of posting on Clinicaltrials.gov

## TABLE OF CONTENTS

| TITLE PAGE | 1 |
|---|---|
| TABLE OF CONTENTS | 2 |
| LIST OF IN-TEXT TABLES AND FIGURES | 3 |
| LIST OF ABBREVIATIONS | 4 |
| 1. INTRODUCTION | 6 |
| 2. STUDY OBJECTIVES | 6 |
| 3. STUDY ENDPOINTS | 6 |
| 4. STUDY DESIGN | 7 |
| 5. SAMPLE SIZE JUSTIFICATION | 8 |
| 6. STUDY TREATMENTS | 9 |
| 7. DEFINITIONS OF POPULATIONS | 10 |
| 7.1. All Subjects Population | 10 |
| 7.2. Safety Population | 10 |
| 7.3. Pharmacokinetic Population | 10 |
| 8. STATISTICAL METHODOLOGY | 10 |
| 8.1. General | 10 |
| 8.1.1. Handling of Data Quality Issues Due to Coronavirus Disease 2019 an Restrictions | |
| 8.1.2. Calculation of the Summary Statistics | 12 |
| 8.1.3. Triplicate Readings | 12 |
| 8.1.4. Repeat and Unscheduled Readings | 13 |
| 8.2. Subject Disposition and Population Assignment | |
| 8.3. Screening Demographics and Baseline Characteristics | 13 |
| 8.4. Prior and Concomitant Medication | 13 |
| 8.5. Pharmacokinetic Assessments | 13 |
| 8.5.1. Pharmacokinetic Analysis | 13 |
| 8.5.2. Presentation of Pharmacokinetic Data | 16 |
| 8.5.3. Pharmacokinetic Statistical Methodology | 17 |
| 8.6. Safety and Tolerability Assessments | 18 |
| 8.6.1. Adverse Events | |
| 8.6.2. Clinical Laboratory Parameters | 20 |
| 8.6.3. Vital Signs Parameters | 20 |

| 8.6.4. 12-lead Electrocardiogram Parameters | 20 |
|--------------------------------------------------------------|----|
| 8.6.5. Other Assessments | 20 |
| 8.6.6. Safety and Tolerability Statistical Methodology | 21 |
| 9. INTERIM ANALYSES | 21 |
| 10. SIGNIFICANT CHANGES FROM THE PROTOCOL-SPECIFIED ANALYSES | 21 |
| 11. REFERENCES | 21 |
| 12. APPENDICES | 22 |
| Appendix 1: Document History | 22 |
| LIST OF IN-TEXT TABLES AND FIGURES | |
| Table 1: Presentation of Study Treatments in TFLs | 9 |
| Table 2: Presentation of Study Treatment Sequences in TFLs | 9 |
| Figure 1: Study Schematic | 8 |

#### LIST OF ABBREVIATIONS

Abbreviations pertain to the statistical analysis plan (SAP) only (not the tables, figures, and listings [TFLs]).

%AUC<sub>extrap</sub> percentage of area under the plasma concentration-time curve due to

extrapolation from the last quantifiable concentration to infinity

ADaM Analysis Data Model

AE adverse event

AUC area under the concentration-time curve

AUC<sub>inf</sub> area under the plasma concentration-time curve from time zero

extrapolated to infinity

AUC<sub>last</sub> area under the plasma concentration-time curve from time zero to the

last quantifiable concentration

BLQ below the limit of quantification

CDISC Clinical Data Interchange Standards Consortium

CDER Center for Drug Evaluation and Research

CI confidence interval

CTCAE Common Terminology Criteria for Adverse Events

CL/F apparent total clearance

C<sub>max</sub> maximum observed plasma concentration

COVID-19 coronavirus disease 2019
CRU clinical research unit
CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

CV coefficient of variation
DMP data management plan
ECG electrocardiogram
EOS end of study

eCRF electronic case report form
GLSM geometric least square means

ICF informed consent form

ICH International Council for/Conference on Harmonisation

 $\lambda_z$  apparent terminal elimination rate constant

 $\lambda_z$  Lower start of exponential fit

 $\lambda_z N$  number of data points included in the log-linear regression

 $\lambda_z$  Span Ratio time period over which lambda z was determined as a ratio of apparent

terminal elimination half-life

 $\lambda_z$  Upper end of exponential fit

LLOQ lower limit of quantification

ln natural log

LSM least squares mean

MedDRA Medical Dictionary for Regulatory Activities

NA not applicable
NC not calculated
PK pharmacokinetic(s)

R<sup>2</sup>-adj adjusted coefficient for determination of exponential fit

SAP statistical analysis plan SD standard deviation

SDV source document verification

 $t_{1/2}$  apparent terminal elimination half-life TEAE treatment-emergent adverse event

TFL table, figure, and listing

 $t_{last}$  time of the last quantifiable plasma concentration  $t_{max}$  time of the maximum observed plasma concentration  $V_z/F$  apparent volume of distribution during the terminal phase

WHODrug World Health Organization Drug Dictionary

#### 1. INTRODUCTION

This SAP has been developed after review of the clinical study protocol (Final Version 1.0) dated 18 February 2022) and electronic case report form (eCRF).

This SAP describes the planned analysis of the pharmacokinetic (PK), safety, and tolerability data from this study. A detailed description of the planned TFLs to be presented in the clinical study report (CSR) is provided in the accompanying TFL shells document.

In general, the analyses are based on information from the protocol, unless they have been modified by agreement with Amgen Inc. A limited amount of information about this study (eg, objectives, study design) is given to help the reader's interpretation.

This SAP must be finalized prior to the lock of the clinical database. Additionally, the SAP and TFL shells should be finalized prior to any programming activities commencing.

This SAP supersedes any statistical considerations identified in the protocol; where considerations are substantially different, they will be so identified. If additional analyses are required to supplement the planned analyses described in this SAP, they may be performed and will be identified accordingly in the CSR. Any substantial deviations from this SAP will be agreed with Amgen Inc. and identified in the CSR.

This SAP is written with consideration of the recommendations outlined in the International Conference on Harmonisation (ICH) E3 guideline Structure and Content of Clinical Study Reports, ICH E8 guideline General Considerations for Clinical Trials, ICH E9 guideline Statistical Principles for Clinical Trials. 1,2,3

The document history is presented in Appendix 1.

#### 2. STUDY OBJECTIVES

The primary objective of the study is:

• to compare the PK of 240 mg sotorasib administered orally as 1 x 240 mg tablet under fasted conditions to 240 mg sotorasib administered orally as 2 x 120 mg tablets under fasted conditions.

The secondary objectives of the study are:

- to evaluate the PK of 240 mg sotorasib administered orally as 1 x 240 mg tablet with a high-fat meal
- to evaluate the safety and tolerability of 240 mg sotorasib administered orally as 1 x 240 mg tablet and 2 x 120 mg tablets.

#### 3. STUDY ENDPOINTS

The primary endpoints of the study are sotorasib PK parameters in Period 1 and Period 2:

- maximum observed plasma concentration (C<sub>max</sub>)
- area under the plasma concentration-time curve (AUC) from time zero to the last quantifiable concentration (AUC<sub>last</sub>)
- area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC<sub>inf</sub>).

The secondary endpoints of the study are:

- adverse events (AE)
- clinical laboratory tests
- 12-lead electrocardiograms (ECGs)
- vital signs
- sotorasib PK parameters in Period 3: C<sub>max</sub>, AUC<sub>last</sub>, AUC<sub>inf</sub>.

#### 4. STUDY DESIGN

This will be an open-label, multi-center (United States), crossover, 3-period study. Groups 1 and 2 will enroll approximately 146 healthy male and healthy female subjects for a duration of at least 2 periods. Approximately 14 out of the 146 (to ensure 12 evaluable subjects) will remain on study for an additional third period. Periods 1 and 2 will comprise the bioequivalence portion of the study where subjects will receive a single oral dose of 240 mg sotorasib administered as 1 x 240 mg tablet (test) and a single oral dose of 240 mg sotorasib administered as 2 x 120 mg tablets (reference) under fasted conditions in the order specified by their assigned group. Period 3 will be the fed portion of the study where a subset of subjects will receive an additional 240 mg sotorasib dose administered as 1 x 240 mg tablet with a high-fat meal to evaluate the PK of sotorasib administered as a 240 mg tablet under fed conditions.

After informed consent is obtained, potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the first dose administration. Subjects will be admitted into the Clinical Research Unit (CRU) on Day -1 and be confined to the CRU until discharge on Day 6 (for subjects enrolled only in Period 1 and Period 2) or Day 9 (for subjects enrolled in all 3 periods). On Day 1, subjects will be randomized to Group 1 or Group 2. Each subject will receive 1 administration of 240 mg sotorasib administered orally under fasted condition as 1 x 240 mg tablet (Treatment A) and 1 administration of 240 mg sotorasib administered orally under fasted condition as 2 x 120 mg tablets (Treatment B) in either Period 1 or Period 2. On Day 7, approximately 14 subjects in either Group 1 or Group 2 will proceed to Period 3 and receive 1 additional administration of 240 mg sotorasib administered orally as 1 x 240 mg tablet with a high-fat meal (Treatment C).

| | 7 11 | | | |
|---|--------|--------|------|-----|
| I | abcorp | Study: | 8471 | 134 |

SAP

| Group | Period 1 (Day 1) | Period 2 (Day 4) | Period 3 (Day 7) |
|---|---|---|---|
| 1 | Treatment A | Treatment B | Treatment C (approximately 14 |
| 2 | Treatment B | Treatment A | subjects from Group 1 or<br>Group 2) |

An overview of the study design is shown in Figure 1.

Figure 1:Study Schematic



The total duration of study participation for each subject (from Screening through end of study [EOS]) is anticipated to be approximately 5 weeks.

The start of the study is defined as the date the first enrolled subject signs an Informed Consent Form (ICF). The point of enrollment occurs at the time of subject number allocation. The end of the study is defined as the date of the last subject's last assessment (scheduled or unscheduled).

#### 5. SAMPLE SIZE JUSTIFICATION

This study will require at least 132 subjects completing Periods 1 and 2 of the study to establish equivalence between 2 treatments with 90% power. This test is based on a 2-sided ratio of means test for a 2 x 2 crossover design for continuous data with significance level 5%. The ratio of means between test and reference under the alternative hypothesis is 0.95. This test assumes lower and upper equivalence limits of 0.8 and 1.25, respectively, and root mean squared error of the log ratio equal to 0.472. Assuming approximately 10% drop-out rate, approximately 146 subjects (73 subjects per treatment) will be enrolled in this study. In

Period 3, approximately 14 subjects planned for food-effect inferential analysis is based on common practice for studies of similar nature and not based on power calculations.

#### 6. STUDY TREATMENTS

The study treatment names, abbreviations, and ordering to be used in the TFLs are presented in Table 1.

Table 1: Presentation of Study Treatments in TFLs

| Treatments | Abbreviation | Order in TFLs |
|---|---|---|
| one administration of 240 mg sotorasib administered orally as 1 x 240 mg tablets | Treatment A | 1 |
| one administration of 240 mg sotorasib administered orally as 2 x 120 mg tablets | Treatment B | 2 |
| one administration of 240 mg sotorasib administered orally as 1 x 240 mg tablets with a high-fat meal | Treatment C | 3 |

The study treatment sequence names, abbreviations, and ordering to be used in the TFLs are presented in Table 2.

Table 2: Presentation of Study Treatment Sequences in TFLs

## For all subjects:

| Study Treatment Sequence | Abbreviation | Order in TFLs |
|---|---|---|
| one administration of 240 mg sotorasib administered orally as 1 x 240 mg tablets on Period 1 (Day 1) and one administration of 240 mg sotorasib administered orally as 2 x 120 mg tablets on Period 2 (Day 4) | Sequence AB | 1 |
| one administration of 240 mg sotorasib administered orally as 2 x 120 mg tablets on Period 1 (Day 1) and one administration of 240 mg sotorasib administered orally as 1 x 240 mg tablets on Period 2 (Day 4) | Sequence BA | 2 |

#### For the 14 subjects attending all 3 periods:

| Study Treatment Sequence | Abbreviation | Order in TFLs |
|---|---|---|
| one administration of 240 mg sotorasib administered orally as 1 x 240 mg tablets on Period 1 (Day 1) and one administration of 240 mg sotorasib administered orally as 2 x 120 mg tablets on Period 2 (Day 4) and one administration of 240 mg sotorasib administered orally as 1 x 240 mg tablets with a high-fat meal (Day 7) | Sequence<br>ABC | 1 |
| one administration of 240 mg sotorasib administered orally as 2 x 120 mg tablets on Period 1 (Day 1) and one administration of 240 mg sotorasib administered orally as 1 x 240 mg tablets on Period 2 (Day 4) and one administration of 240 mg sotorasib administered orally as 1 x 240 mg tablets with a high-fat meal (Day 7) | Sequence<br>BAC | 2 |

The summaries will be based on planned treatment sequences and listings will be based on actual treatment sequences (eg, if subject was assigned to receive placebo in Period 1 and active treatment in Period 2 (sequence [A/B]) but was wrongfully dosed with active treatment in Period 1 and discontinued before start of Period 2, they would be summarized under 'A/B' treatment sequence and listed under 'B' treatment sequence).

#### 7. DEFINITIONS OF POPULATIONS

Any protocol deviations, including those due to coronavirus disease 2019 (COVID-19) and related restrictions (see Section 8.1.1), will be considered prior to database lock for their importance and taken into consideration when assigning subjects to populations.

#### 7.1. All Subjects Population

The all subjects population will include all subjects who signed the ICF and had any study assessment recorded in the database per the protocol.

#### 7.2. Safety Population

The safety population will include all subjects who received at least 1 dose of sotorasib.

#### 7.3. Pharmacokinetic Population

The PK population will include all subjects who received at least 1 dose of sotorasib and have evaluable PK data. A subject may be excluded from the PK summary statistics and statistical analysis if the subject has an adverse events of vomiting that occurs at or before 2 times median time to maximum concentration or diarrhea within 24 hours of dosing.

#### 8. STATISTICAL METHODOLOGY

#### 8.1. General

Listings will be provided for all data captured in the database, with the exception of medical history. Listings will include all subjects assigned to the all subjects population and include

data up to the point of study completion or discontinuation. Subjects are generally considered to have completed the study if they complete the scheduled end of study visit (rather than early termination visit). Any subject who discontinues the study will be identified accordingly in the listings. Summaries and statistical analyses will include the subjects assigned to the relevant population based on data type.

Data analysis will be performed using the SAS® statistical software package Version 9.4 (or higher if a new version is issued during the study).

Analysis Data Model (ADaM) datasets will be prepared using Clinical Data Interchange Standards Consortium (CDISC) ADaM Version 2.1 (or higher if a new version is issued during the study) and CDISC ADaM Implementation Guide Version 1.1 (or higher if a new version is issued during the study). Pinnacle 21 Community Version 4.0.0 (or higher if a new version is issued during the study) will be utilized to ensure compliance with CDISC standards.

Where reference is made to 'valid' data, this refers to non-missing data which meet the predetermined criteria (eg, are not flagged for exclusion).

Where reference is made to 'all calculations', this includes, but is not limited to, summary statistics, statistical analyses, baseline derivation, changes from baseline, percentage changes from baseline, and any parameter derivations.

All figures will be produced on linear-linear or discrete-linear scales, as applicable, unless specifically stated otherwise.

# 8.1.1. Handling of Data Quality Issues Due to Coronavirus Disease 2019 and Related Restrictions

Due to COVID-19 and related restrictions, there is a high risk for impact to data integrity, with the recognized potential for:

- Missed visits, caused by, for example:
  - Subject unable to travel to site due to restrictions, the need to quarantine, or COVID-19 infection
  - o Subject unwilling to go to site due to fear of COVID-19 infection
  - o Site postponing subject's visit due to investigator not being available (eg, if they have been dispatched to hospital handling COVID19 infections)
- Site unable to replenish supply of investigational product
- Incomplete data entry by sites due to limited resources to support study or no access to source documents or to eCRF
- Outstanding source document verification (SDV) due to sponsor or country restrictions on remote SDV, or no or limited access to site(s) for on-site visits

#### • Unanswered queries

At the time of the reporting of the study results, all protocol deviations due to COVID-19 or related restriction will be assessed for their severity and impact on the analyses. If needed, appropriate statistical methods will be applied as a mitigating action (eg, data might be categorized into 2 analysis groups, with and without COVID-19 and related restrictions impact); however, this will exclude any imputations of the missing values. Any mitigating actions will be agreed with Amgen Inc. in advance and identified in the CSR.

#### 8.1.2. Calculation of the Summary Statistics

For continuous data the following rules will be applied:

- Missing values will not be imputed, unless specifically stated otherwise.
- Unrounded data will be used in the calculation of summary statistics.
- If the number of subjects with valid observations (n) <3, summary statistics will not be calculated, with the exception of n, minimum, and maximum.
- In general, as early termination data are not associated with any scheduled timepoint, they will be excluded from all calculations of summary statistics and statistical analyses. Exceptions may be made where justified.

For categorical data the following rules will be applied:

- For ordered categorical data (eg, AE severity), all categories between the possible minimum and maximum categories will be included, even if n = 0 for a given category.
- For non-ordered categorical data (eg, race), only those categories for which there is at least 1 subject represented will be included; unless specifically stated otherwise.
- Missing values will not be imputed, unless specifically stated otherwise. A 'missing' category will be included for any parameter for which information is missing. This will ensure that the population size totals are consistent across different parameters.

#### 8.1.3. Triplicate Readings

For 12-lead electrocardiogram (ECG) data only, where triplicate readings are taken, the mean of triplicate readings will replace the separate individual triplicate readings in all calculations.

In case of incomplete triplicate readings (eg, only 2 out of 3 readings were recorded), the mean and/or medians will be calculated, as appropriate, based on the number of readings available.

#### 8.1.4. Repeat and Unscheduled Readings

For vital signs and 12-lead ECG data only, any predose value recorded in addition to the original value or a postdose value recorded within 15 minutes of the original value will be defined as a repeat value; any postdose value recorded more than 15 minutes after the original value will be defined as an unscheduled value. For all other data types (eg, laboratory parameters), any value recorded in addition to the original value will be defined as an unscheduled value.

The original value will be replaced by the last associated repeat value in all calculations.

As unscheduled values are not associated with any scheduled timepoint, they will be excluded from all calculations.

#### 8.2. Subject Disposition and Population Assignment

Subject disposition and population assignment will be listed.

A summary table by treatment will be provided, based on the safety population.

#### 8.3. Screening Demographics and Baseline Characteristics

The screening demographics and baseline characteristics including sex, age, race, ethnicity, height, body weight, and body mass index will be listed.

A summary table by treatment will be provided, based on the safety population.

#### 8.4. Prior and Concomitant Medication

Prior medication will be defined as medication that ends prior to first dosing. Concomitant medication will be defined as medication that starts during or after first dosing or starts but does not end prior to first dosing.

Prior and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHODrug) Global, Format B3, Version September 2020 (or later if a new version is issued during the study; see the data management plan [DMP] for more details). Prior and concomitant medications will be listed.

#### 8.5. Pharmacokinetic Assessments

#### 8.5.1. Pharmacokinetic Analysis

The following PK parameters will be determined on Day 1, Day 4, and Day 7, data permitting, from the plasma concentrations of sotorasib using noncompartmental methods in validated installation of Phoenix WinNonlin (Certara, Version 8.1.1 or higher):


| SAP | | | |
|---------|--------|------|-----|
| Labcorp | Study: | 8471 | 134 |

CAD

| Parameter | Unitsa | Definition |
|---|---|---|
| AUC <sub>last</sub> | h*ng/mL | area under the plasma concentration-time curve from time zero to the last quantifiable concentration <sup>b</sup> |
| $AUC_{\mathrm{inf}}$ | h*ng/mL | area under the plasma concentration-time curve from time zero extrapolated to infinity <sup>c</sup> |
| $C_{\text{max}}$ | ng/mL | maximum observed plasma concentration |
| $t_{\text{max}}$ | h | time of the maximum observed plasma concentration |
| $t_{last}$ | h | time of the last quantifiable plasma concentration |
| $t_{1/2}$ | h | apparent terminal elimination half-life |
| CL/F | L/h | apparent total clearance |
| $V_z/F$ | L | apparent volume of distribution during the terminal phase |

<sup>&</sup>lt;sup>a</sup> Units are based on concentration units (provided by the bioanalytical lab or preferred units for presentation of PK parameters) and dose units used in the study.

Additional PK parameters may be determined where appropriate.

Pharmacokinetic analysis will be carried out where possible using actual dose administered (mg) and actual postdose blood sampling times. If an actual time is missing, nominal times may be used with sponsor's approval.

The parameters C<sub>max</sub>, t<sub>last</sub>, and t<sub>max</sub> will be obtained directly from the concentration-time profiles.

For multiple peaks, the highest postdose concentration will be reported as C<sub>max</sub>. In the case that multiple peaks are of equal magnitude, the earliest t<sub>max</sub> will be reported.

#### 8.5.1.1. Criteria for the Calculation of Apparent Terminal Elimination Rate Constant and Half-life

The start of the terminal elimination phase for each subject will be defined by visual inspection and generally will be the first point at which there is no systematic deviation from the log-linear decline in concentrations.

The apparent terminal elimination rate constant ( $\lambda_z$ ) will only be calculated when a reliable estimate can be obtained using at least 3 data points, preferably not including C<sub>max</sub>, and the adjusted coefficient for determination of exponential fit ( $R^2$ -adj) of the regression line is  $\geq 0.8$ . Parameters requiring  $\lambda_z$  for their calculation (eg, AUC<sub>inf</sub>,  $t_{1/2}$ , CL/F, and  $V_z/F$ ) will only be calculated if the  $R^2$ -adj value of the regression line is  $\geq 0.8$ .

The following regression-related diagnostic PK parameters will be determined, when possible:


b Area under the plasma concentration-time curve will be calculated using the linear trapezoidal rule.

<sup>&</sup>lt;sup>c</sup> Based on the last observed quantifiable concentration.

| Parameter | Units | Definition |
|---|---|---|
| %AUC <sub>extrap</sub> | % | percentage of area under the plasma concentration-time curve due to extrapolation from the last quantifiable concentration to infinity |
| $\lambda_z$ | 1/h | apparent terminal elimination rate constant |
| $\lambda_z$ Upper | h | end of exponential fit |
| $\lambda_z$ Lower | h | start of exponential fit |
| $\lambda_zN$ | NA | number of data points included in the log-linear regression |
| $\lambda_z$ Span Ratio | NA | time period over which $\lambda_z$ was determined as a ratio of $t_{1/2}$ |
| R <sup>2</sup> -adj | NA | adjusted coefficient for determination of exponential fit |

Where possible, the span of time used in the determination of  $\lambda_z$  (ie, the difference between  $\lambda_z$  Upper and  $\lambda_z$  Lower) should be  $\geq 2$  half-lives. If the  $\lambda_z$  span ratio is  $\leq 2$ , the robustness of the  $t_{1/2}$  values will be discussed in the CSR.

# 8.5.1.2. Criteria for Calculation and Reporting of Area Under the Concentration-time Curve

The minimum requirement for the calculation of AUC will be the inclusion of at least 3 consecutive concentrations above the lower limit of quantification (LLOQ). If there are only 3 consecutive concentrations, at least 1 should follow  $C_{max}$ .

If the extrapolated area is >20%, AUC<sub>inf</sub> (and derived parameters) will be flagged and may be excluded from the summary statistics and statistical analysis at the discretion of the sponsor or pharmacokineticist.

If AUC<sub>inf</sub> cannot be determined reliably for all subjects and/or treatments, an alternative AUC measure, such as AUC to a fixed timepoint or AUC<sub>last</sub>, may be used in the statistical analysis upon sponsor approval.

# 8.5.1.3. Criteria for Handling Below the Limit of Quantification or Missing Concentrations for Pharmacokinetic Analysis

Plasma concentrations below the limit of quantification (BLQ) will be assigned a value of 0 before the first measurable concentration and thereafter BLQs will be treated as missing. The following rules apply to the specific situations defined below:

- If an entire concentration-time profile is BLQ, it will be excluded from PK analysis.
- Where 2 or more consecutive concentrations are BLQ at the end of a profile, the profile will be deemed to have terminated and any further quantifiable concentrations will be set to missing for the calculation of the PK parameters, unless they are considered to be a true characteristic of the profile of the drug.
- If a predose plasma concentration is missing, it will be set to 0 by default within Phoenix WinNonlin.

#### 8.5.1.4. Treatment of Outliers in Pharmacokinetic Analysis

If a value is considered to be anomalous due to being inconsistent with the expected PK profile, it may be appropriate to exclude the value from the PK analysis. However, the exclusion of any data must have strong justification and will be documented in the CSR.

Any quantifiable predose concentration value in the first treatment period will be considered anomalous and set to missing for the PK analysis. This will be set to 0 by default in Phoenix WinNonlin.

If the predose concentration is >5% of  $C_{max}$  in the second or third treatment periods, all PK concentration and parameter data will be flagged and reported, but excluded from the summary statistics and statistical analysis for that period.

#### 8.5.2. Presentation of Pharmacokinetic Data

If the actual time of sample collection deviates from the nominal time by more than  $\pm 10\%$ , the plasma concentration will be flagged and excluded from the summary statistics.

Individual concentrations deemed to be anomalous will be flagged in the listings and excluded from the summary statistics.

For plasma concentration data the following rules will apply:

- Values that are BLQ will be set to 0 for the calculation of summary statistics.
- If the embedded BLQ value is considered anomalous within the concentration-time profile, this value will be excluded from the summary statistics.
- Where there is NR, these will be set to missing.
- If there are less than three values in the data series, only the min, max and N will be presented. The other summary statistics will be denoted as not calculated (NC). BLQ is considered a value.
- If the values are BLQ, then the arithmetic mean, arithmetic SD, median, min and max will be presented as 0 and the geometric mean and geometric coefficient of variation (CV%) will be denoted as NC.
- Arithmetic mean or median values that are BLQ will be presented as 0, and the geometric mean and geometric CV% will be denoted as NC.

For PK parameters the following rules will apply:

- For the calculation of summary statistics of PK parameters, all non-reportable and NC values in a data series will be set to missing.
- AUC $_{inf}$  and AUC $_{last}$  will be set to NC if they were calculated using fewer than three concentrations, and/or three concentrations if the last is  $C_{max}$ .

• Geometric mean and coefficient of variation will not be calculated for  $t_{last}$  or  $t_{max}$ .

#### 8.5.3. Pharmacokinetic Statistical Methodology

All PK concentrations and parameters will be listed.

Summary tables, mean (+ standard deviation [SD]) figures, overlaying individual figures, and individual figures by treatment and time postdose will be provided for plasma PK concentrations. All figures will be produced on both linear and semi-logarithmic scales.

Summary tables by treatment will be provided for all PK parameters, with the exception of regression-related PK parameters.

#### Bioequivalence:

A statistical analysis will be conducted to investigate the bioequivalence of 240 mg sotorasib administered orally as 1 x 240 mg tablets (test) to 240 mg sotorasib administered orally as 2 x 120 mg tablets (reference) for  $AUC_{last}$ ,  $AUC_{infb}$  and  $C_{max}$ . Data from the entire study population will be used for this analysis.

The natural log (ln)-transformed<sup>4</sup> PK parameters will be analyzed using a mixed model.<sup>5</sup> The model will include treatment, period, and sequence as fixed effect and subject nested within sequence as a random effect.

For AUC<sub>last</sub>, AUC<sub>inf</sub> and C<sub>max</sub> separately, the least squares mean (LSM) for each treatment, difference in LSMs between the test and reference treatments, and corresponding 90% confidence interval (CI) will be calculated; these values will then be back-transformed to give the geometric least square mean (GLSM), ratio of GLSMs, and corresponding 90% CI.

Additionally, the pooled estimate (across all treatments) of the within-subject CV will be calculated, and residual plots will be produced to assess the adequacy of the model(s) fitted.

It will be concluded that the test treatment is bioequivalent to the reference treatment if, for  $C_{max}$  and AUCs, the 90% CI for the ratio of GLSMs is completely contained within the predefined interval of (0.8000, 1.2500).<sup>6</sup> This procedure is equivalent to Schuirmann's<sup>7</sup> two one-sided tests at the 0.05 level of significance.

Examples of the SAS code that will be used are as follows:



Final Version 1.0, 02June2022

Page 17 of 22 ST-AD-031 Version 02

#### **Food Effect:**

A statistical analysis will be conducted to investigate the food effect for 240 mg sotorasib administered orally as 1 x 240 mg tablets under fed condition (test) to 240 mg sotorasib administered orally as 1 x 240 mg tablets under fasted condition (reference) for  $AUC_{last}$ ,  $AUC_{inf}$  and  $C_{max}$ . Data from 14 subjects who are enrolled in Period 3 will be used for this analysis.

The natural log (ln)-transformed<sup>4</sup> PK parameters will be analyzed using a mixed model.<sup>5</sup> The model will include treatment as fixed effect and subject as a random effect.

For  $AUC_{last}$ ,  $AUC_{infb}$  and  $C_{max}$  separately, the least squares mean (LSM) for each treatment, difference in LSMs between the test and reference, and corresponding 90% confidence interval (CI) will be calculated; these values will then be backtransformed to give the geometric least square mean (GLSM), ratio of GLSMs, and corresponding 90% CI.

Additionally, the pooled estimate (across all treatments) of the within-subject CV will be calculated, and residual plots will be produced to assess the adequacy of the model(s) fitted.

Examples of the SAS code that will be used are as follows:



8.6. Safety and Tolerability Assessments

#### 8.6.1. Adverse Events

All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 24.1 (or higher if a new version is issued during the study; see the DMP for more details). All AEs will be assigned a severity grade using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (or higher if a new version is issued during the study; see the protocol for more details).

A treatment-emergent adverse event (TEAE) will be defined as an AE that starts during or after dosing, or starts prior to dosing and increases in severity after dosing within each period.

A treatment-related TEAE will be defined as a TEAE with a relationship related to the study treatment, as determined by the investigator.


All AEs will be listed. In addition to the data recorded in the database, the listings will include derived onset time and duration. Onset time will be calculated from the time of dosing for TEAEs only.

The frequency of subjects with TEAEs and the number of TEAEs will be summarized for the following categories:

- TEAEs (overall, serious, leading to discontinuation, and leading to death) by treatment
- TEAEs by severity and treatment
- Treatment-related TEAEs (overall, serious, leading to discontinuation, and leading to death) by treatment
- Treatment-related TEAEs by severity and treatment

The frequency of subjects will be summarized separately for TEAEs and treatment-related TEAEs by the following:

- System organ class, preferred term, and treatment
- Preferred term and treatment

For the AE data the following rules will apply:

- For the derivation of treatment-emergent status (applicable to all AEs): If the start date/time of an AE is incomplete or missing, an AE will be assumed to not be a TEAE, unless the incomplete start date/time or the end date/time indicates an AE started after dosing.
- For the derivation of treatment-related status (applicable to TEAEs only): If the study treatment relationship for a TEAE is missing, a TEAE will be assumed to not be a treatment-related TEAE.
- For the derivation of onset time (applicable to TEAEs only): If the start date/time of a TEAE is missing, onset time will not be calculated. If the start date/time of a TEAE is incomplete, where possible, the minimum possible onset time will be calculated and presented in '≥DD:HH:MM' format (eg, if the date/time of dosing is 01MAY2019/08:00 and recorded start date/time of a TEAE is 03MAY2019, then the minimum possible onset time will be calculated by assuming a TEAE started at the first hour and minute of 03MAY2019 [03MAY2019/00:00], thus will be presented as onset time ≥01:16:00 in the listing). If the start date of a TEAE is the same as the date of dosing but the start time of a TEAE is missing, an onset time will be presented as '≥00:00:01'. Any clock changes will be accounted for in the derivation.
- For the derivation of duration (applicable to all AEs): If the end date/time of an AE is missing, duration will not be calculated. If the start or end date/time of an AE is incomplete, where possible, the maximum possible duration will be calculated and

presented in '≤DD:HH:MM' format (eg, if the start of an AE date/time is 01MAY2019/08:00 and its recorded end date/time is 03MAY2019, then the maximum possible duration will be calculated by assuming an AE ended at the last hour and minute of 03MAY2019 [03MAY2019/23:59], thus will be presented as duration ≤02:15:59 in the listing). Any clock changes will be accounted for in the derivation.

- For the calculation of TEAE summary statistics: If the severity of a TEAE is missing, that TEAE will be counted under the 'missing' category.
- For the calculation of TEAE summary statistics: If a subject experienced multiple TEAEs with the same preferred term for the same treatment, this will be counted as 1 TEAE for that treatment under the maximum severity recorded.

#### 8.6.2. Clinical Laboratory Parameters

All clinical laboratory parameters, will be listed, as applicable; any value outside the clinical reference range will be flagged. Separate listings will be provided for any parameter for which there is any individual subject value outside the respective clinical reference range.

Summary tables by treatment and timepoint will be provided for clinical chemistry and hematology parameters.

Values recorded as  $\langle x, \leq x, \rangle x$ , or  $\geq x$  will be displayed in the listings as recorded. For the derivation of listing flags, all calculations, and presentation in the figures,  $\langle x \rangle x$  and  $\leq x \rangle x$  will be set to 0, whereas  $\geq x \rangle x$  and  $\geq x \rangle x$  values will be set to x.

### 8.6.3. Vital Signs Parameters

All vital signs parameters, will be listed, as applicable; any value outside the clinical reference range will be flagged.

Summary tables by treatment and timepoint will be provided by treatment group for all vital signs parameters as applicable.

#### 8.6.4. 12-lead Electrocardiogram Parameters

All 12-lead ECG parameters will be listed; any value outside the clinical reference range will be flagged.

Summary tables by treatment and timepoint will be provided for all 12-lead ECG parameters.

#### 8.6.5. Other Assessments

Medical history will not be listed.

All other safety and tolerability assessments not detailed in the above sections will be listed only.

#### 8.6.6. Safety and Tolerability Statistical Methodology

No inferential statistical analyses are planned.

#### 9. INTERIM ANALYSES

No interim analyses are planned.

#### 10. SIGNIFICANT CHANGES FROM THE PROTOCOL-SPECIFIED ANALYSES

There were no significant changes from the protocol-specified analyses.

#### 11. REFERENCES

- 1. ICH. ICH Harmonised Tripartite Guideline: Structure and content of clinical study reports (E3). 30 November 1995.
- 2. ICH. ICH Harmonised Tripartite Guideline: General considerations for clinical trials (E8). 17 July 1997.
- 3. ICH. ICH Harmonised Tripartite Guideline: Statistical principles for clinical trials (E9). 5 February 1998.
- 4. Keene ON. The log transformation is special. Stat Med. 1995;14(8):811-819.
- 5. Brown H, Prescott R. Applied Mixed Models in Medicine. Chichester: John Wiley & Sons, 1999.
- 6. Statistical Approaches to Establishing Bioequivalence. Rockville, MD: US Dept of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER); January 2001.
- 7. Schuirmann DJ. A comparison of the two one sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987;15(6):657-680.


SAP CONFIDENTIAL Labcorp Study: 8471134 Protocol Reference: 20210088

## 12. APPENDICES

# **Appendix 1: Document History**

| Status and Version | <b>Date of Change</b> | Summary/Reason for Changes |
|-------------------------|-----------------------|----------------------------|
| First Draft Version 1.0 | NA | NA; the first version. |

 $\overline{NA} = not applicable$ 

# Statistical Analysis Plan (SAP) Approval Form

#### Type of Approval (select one): SAP

| Sponsor Name: | Amgen, Inc. | | |
|---|---|---|---|
| Sponsor<br>Protocol<br>/CIP ID: | 20210088 | Covance<br>Study ID: | 8471134 |
| SAP text filenam e: | Amgen510_20210088_SAP_02June 2022_Final.pdf | TFL shells filename: | Amgen510_20210088_TFL_02June 2022_Final.pdf |
| Version: | 1.0 | Date: | 02June2022 |

#### **Covance Approval:**

Lead Statistician



#### **Sponsor Approval:**

By signing below when the statistical analysis plan (SAP) is considered final, the signatories agree to the analyses to be performed for this study and to the format of the associated tables, figures, and listings (TFLs). Once the SAP has been signed, programming of the Analysis Dataset Model (ADaM) datasets and TFLs based on these documents can proceed. Any modifications to the SAP text and TFL shells made after signing may result in a work-scope change.



Please scan/email completed form(s) to the Lead Statistician listed below:

| Printed Name/Title: | , Biostatistician |
|---------------------|-------------------|
| Email: | |

# 16.1.9.2. Quality Tolerance Limits Definitions

| Parameter | Justification for Parameter | Unit Tolerance |
|---|---|---|
| Minimum number of evaluable subjects needed. | A shortfall in the overall number of subjects could have a significant impact on interpretation of the primary endpoint because of limited/insufficient exposure. | N: 132 |

CONFIDENTIAL

Protocol Reference: 20210088

Final 